CLINICAL TRIAL: NCT04983940
Title: Patient Satisfaction After Switching to Oral Testosterone Undecanoate in Men Currently on Testosterone Therapy
Brief Title: Patient Satisfaction After Switching to Oral Testosterone Undecanoate
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Clarus Therapeutics, Inc. (Industry)
Responsible Party: Principal Investigator, Ranjith Ramasamy, MD, Associate Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20200971
Record Dates: First submitted 2021-07-20; First posted 2021-07-30 (Actual); Results first posted 2023-12-14 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-11

CONDITIONS: Testosterone Deficiency
MeSH Terms: interventions — Testosterone Propionate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Jatenzo Arm (Experimental): Participants in this group will receive Jatenzo for 26 consecutive weeks.
  Interventions: Drug: Jatenzo

INTERVENTIONS:
Drug: Jatenzo — 237 mg soft gel capsule taken twice a day by mouth with food.

SUMMARY:
The purpose of this research study is to evaluate patient satisfaction with an oral testosterone agent, Jatenzo, compared to other forms of testosterone therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign and date the study consent form(s) which have been approved by an Institutional Review Board (IRB). Written consent must be obtained prior to the initiation of any study procedures.
2. Males between 18 and 65 years of age.
3. Documented diagnosis of testosterone deficiency.
4. Prior treatment with testosterone therapy at the time of enrollment with adequate control of low testosterone symptoms. Serum total testosterone < 300 ng/dL on 2 measurements prior to the initiation of testosterone therapy. Patients must have completed an adequate washout period following prior testosterone therapy (4 weeks for gels and injection based therapies and 16 weeks for subcutaneous pellets).
5. Judged to be in good general health as determined by the principal investigator based upon the results of a medical history, physical examination, vital signs, laboratory profile and a 12-lead electrocardiogram (ECG).

Exclusion Criteria:

1. History of significant sensitivity or allergy to androgens or product excipients.
2. Clinically significant findings in the pre-study examinations including abnormal breast examination requiring follow-up or abnormal ECG.
3. Abnormal prostate digital rectal examination (DRE) with palpable nodule(s) or International Prostate Symptom Score (I-PSS) score > 19 points.
4. Body mass index (BMI) ≥ 40 kg/m2.
5. Clinically significant abnormal laboratory value, in the opinion of the investigator, in serum chemistry, hematology, or urinalysis including but not limited to:

   1. Baseline hemoglobin > 16 g/dL
   2. Hematocrit < 35% or > 50%
6. Poorly controlled blood pressure as defined by Systolic Blood Pressure (SBP) >150 or Diastolic Blood Pressure (DBP) > 90 on two separate measurements
7. Concurrent use of any prohibited medications that can affect testosterone levels or metabolism.
8. History of seizures or convulsions, including febrile, alcohol or drug withdrawal seizures.
9. History of any clinically significant illness, infection, or surgical procedure within 4 weeks prior to study drug administration.
10. History of stroke or myocardial infarction within the past 5 years.
11. History of, or current or suspected, prostate or breast cancer.
12. History of, or current or suspected, pituitary abnormality.
13. History of diagnosed, severe, untreated, obstructive sleep apnea.
14. History of abuse of alcohol or any drug substance in the opinion of the investigator within the previous 2 years.
15. Receipt of any investigational product within 4 weeks or within 5 half-lives prior to the start of treatment.
16. Inability to understand and provide written informed consent for the study.
17. Considered by the investigator or the sponsor-designated physician, for any reason, that the subject is an unsuitable candidate to receive Jatenzo

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2021-06-18 (Actual); Primary Completion 2023-04-06 (Actual); Study Completion 2023-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ranjith Ramasamy, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Jatenzo Arm
Started | 41
Completed | 25
Not Completed | 16
Not completed — Lost to Follow-up | 14
Not completed — Lack of Efficacy | 2

BASELINE CHARACTERISTICS:
Arm/Group | Jatenzo Arm
Number analyzed (Participants) | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.8 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 34
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Patient Satisfaction as Measured by TSQM-9 (Global Satisfaction Domain)
Description: Treatment Satisfaction Questionnaire for Medication (TSQM-9) has three domains (Global, Convenience, and Effectiveness), each with a total score ranging from 0 to 100 with the higher score indicating higher patient satisfaction.
Time Frame: Up to 6 months
Population: Some participants did not complete all of the study visits due to non compliance with the protocol.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Jatenzo Arm
Number analyzed (Participants) | 30
score on a scale
  Baseline | 66.7 [55.3 to 78.1]
  Month 3: number analyzed (Participants) | 27
  Month 3 | 83.1 [76.8 to 89.3]
  Month 6: number analyzed (Participants) | 25
  Month 6 | 83.7 [75.5 to 91.9]

2. Primary Outcome: Hypogonadal Symptoms as Measured by qADAM Questionnaire
Description: Quantitative Androgen Deficiency in the Aging Male (qADAM) has a total score ranges between 10 (most symptomatic) and 50 (least symptomatic).
Time Frame: Up to 6 months
Population: Some participants did not complete all of the study visits due to non compliance with the protocol.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Jatenzo Arm
Number analyzed (Participants) | 30
score on a scale
  Baseline | 36.6 [35.7 to 37.5]
  Month 3: number analyzed (Participants) | 27
  Month 3 | 34.4 [32.9 to 36.0]
  Month 6: number analyzed (Participants) | 25
  Month 6 | 35.5 [33.5 to 37.6]

3. Secondary Outcome: Serum Testosterone Levels
Description: Serum testosterone levels measured in ng/dL analyzed from peripheral venous puncture blood draw
Time Frame: Up to 6 months
Population: Some participants did not complete all of the study visits due to non compliance with the protocol.
Measure: Mean (95% Confidence Interval); unit: ng/dL
Arm/Group | Jatenzo Arm
Number analyzed (Participants) | 30
ng/dL
  Baseline | 200.3 [177.7 to 222.9]
  Month 3: number analyzed (Participants) | 27
  Month 3 | 486.8 [398.9 to 574.7]
  Month 6: number analyzed (Participants) | 24
  Month 6 | 649.3 [504.0 to 794.7]

4. Secondary Outcome: Serum Estradiol Levels
Description: Serum estradiol levels measured in pg/mL analyzed from peripheral venous puncture blood draw.
Time Frame: Up to 6 months
Population: Estradiol was added to the protocol during an amendment after the trial had begun. Some participants did not complete all of the study visits due to non-compliance with the protocol.
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Jatenzo Arm
Number analyzed (Participants) | 23
pg/mL
  Baseline | 14.4 [11 to 17.8]
  Month 3: number analyzed (Participants) | 21
  Month 3 | 21.6 [16.9 to 26.3]
  Month 6: number analyzed (Participants) | 17
  Month 6 | 21.2 [15.8 to 26.7]

5. Secondary Outcome: Hematocrit Levels
Description: Hematocrit levels measured as a percentage analyzed from peripheral venous puncture blood draw.
Time Frame: Up to 6 months
Population: Some participants did not complete all of the study visits due to non-compliance with the protocol.
Measure: Mean (95% Confidence Interval); unit: percentage of hematocrit
Arm/Group | Jatenzo Arm
Number analyzed (Participants) | 30
percentage of hematocrit
  Baseline | 44.9 [43.5 to 46.4]
  Month 3: number analyzed (Participants) | 27
  Month 3 | 45 [43.6 to 46.5]
  Month 6: number analyzed (Participants) | 24
  Month 6 | 45.2 [43.9 to 46.5]

6. Secondary Outcome: PSA Levels Measured in ng/mL
Description: Prostate Specific Antigen (PSA) levels measured in ng/mL analyzed from peripheral venous puncture blood draw.
Time Frame: Up to 6 months
Population: PSA was added to the protocol during an amendment after the trial had begun. Some participants did not complete all of the study visits due to non-compliance with the protocol.
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Jatenzo Arm
Number analyzed (Participants) | 23
ng/mL
  Baseline | 1.06 [0.71 to 1.41]
  Month 3: number analyzed (Participants) | 21
  Month 3 | 1.14 [0.80 to 1.49]
  Month 6: number analyzed (Participants) | 17
  Month 6 | 0.95 [0.53 to 1.37]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Jatenzo Arm
All-Cause Mortality (participants affected / at risk) | 0/41
Serious Adverse Events (participants affected / at risk) | 1/41
Other Adverse Events (participants affected / at risk) | 5/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Jatenzo Arm (N=41)
Chronic Kidney Disease (Renal and urinary disorders) | 1 (1) — Chronic Kidney Disease requiring Kidney Transplant
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Jatenzo Arm (N=41)
Hypertension (Vascular disorders) | 3 (3)
Polycythemia (Blood and lymphatic system disorders) | 1 (1)
Nocturia (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-19): https://cdn.clinicaltrials.gov/large-docs/40/NCT04983940/Prot_SAP_000.pdf